CLINICAL TRIAL: NCT06948929
Title: A Pilot, Single-arm Study on the Efficacy and Safety of the Use of a Synbiotic Formula (SCV09) in Alzheimer's Disease Patients
Brief Title: Synbiotic Formula (SCV09) in Alzheimer's Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024.530
Record Dates: First submitted 2025-04-28; First posted 2025-04-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm intervention only (Experimental): SV09
  1 sachet daily for 6 months
  Interventions: Dietary Supplement: SCV09

INTERVENTIONS:
Dietary Supplement: SCV09 — SCV09 consists of a blend of four probiotic species from the Bifidobacterium and Lactobacillus genera (20 billion CFU in 1 sachet per day), prebiotic compounds including galacto-oligosaccharides, xylo-oligosaccharides and inulin, vitamin B6, B9, B12 and vitamin D.

SUMMARY:
In recent years, emerging studies have revealed the role of gut microbiota in human health and diseases, including AD and other neurodegenerative conditions5. Although the underlying mechanism is still largely unknown, successful therapies targeting the gut-brain axis may serve as indirect evidence of the possible linkage.

This pilot, single-arm study aims to estimate the efficacy and assess the safety profile of the use of a new synbiotic formula (SCV09) in improving dementia-related behaviour in Alzheimer's disease patients, paving the way for a large-scale randomised controlled trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 60-85 with a clinical diagnosis of Alzheimer's disease
* Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) score of ≤20
* Neuropsychiatric Inventory-Questionnaire (NPI-12) ≥10
* Stable medication history for Alzheimer's disease within the past 4 weeks
* Have been taken care by a responsible caregiver who could assist the patient in taking the study products, collecting stool samples and attending the clinical follow-up •-Able to provide informed consent

Exclusion Criteria:

* Concomitant Parkinson's disease and other neurodegenerative conditions affecting activities of daily living
* History of stroke
* History of severe organ failure (including decompensated cirrhosis), renal failure on dialysis, suffering from human immunodeficiency virus infection
* Confirmed active malignancy
* Known operations involving small intestines and large intestines; or history of appendectomy, hysterectomy, and cholecystectomy in last 6 months
* Use of anti-psychotics, antidepressants or sedatives, unless on a stable dose in the last 3 months
* Inability to receive oral fluids
* Use of antibiotics, probiotics or prebiotics in the last 2 weeks
* Intolerance to probiotics or lactose

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory-Questionnaire | 6 months
  Proportion of subjects who have no change or at least a 1 point decrease in Neuropsychiatric Inventory-Questionnaire (NPI-12) score

SECONDARY OUTCOMES:
Activities of Daily Living | 6 months
  Changes in activities of daily living, assessed by Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
HK-MoCA | 6 months
  Changes in Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) score
Gut microbiota composition and functions | 6 months
  Explore the gut microbiota composition and functions from stool sample

CONTACTS AND LOCATIONS:
Overall Officials: Professor Timothy Kwok, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinse University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No